CLINICAL TRIAL: NCT06825403
Title: Olfactory Training in Mild Cognitive Impairment
Acronym: OTMCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Motter (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Motter, Research Scientist, New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00082984; AARG-24-1301387 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Olfactory Training; Olfactory Memory Training; Visual Training; Visual Memory Training; Olfaction; Memory Disorders; Cognitive Disorders; Cognitive Impairment; Mild Cognitive Impairment; Cognitive Training
MeSH Terms: conditions — Cognitive Dysfunction; Anosmia; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either Olfactory Memory Training (OMT) or Visual Memory Training (VMT) by random number generators.
Masking Description: Due to the pilot nature of the study and fundamental differences between OMT and VMT, neither the participants nor research personnel will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olfactory Memory Training (Active Comparator)
  Interventions: Behavioral: Olfactory Memory Training
- Visual Memory Training (Active Comparator)
  Interventions: Behavioral: Visual Memory Training

INTERVENTIONS:
Behavioral: Olfactory Memory Training — Participants will complete 48 OMT sessions at home lasting approximately 10 minutes each over 3 months.
  Arms: Olfactory Memory Training
Behavioral: Visual Memory Training — Participants will complete 48 VMT sessions at home lasting approximately 10 minutes each over 3 months.
  Arms: Visual Memory Training

SUMMARY:
Sense of smell tends to decline in individuals with early Alzheimer's disease, typically earlier than when other senses and thinking abilities begin to decline. Memory for new odors is particularly diminished in these individuals. Existing treatments for AD do not improve these symptoms. A targeted treatment for improving sense of smell, called 'Olfactory Training', has been used to improve sense of smell in people with various forms of smell loss, though it is not known whether it can improve smell abilities and thinking abilities in patients who are at high risk of developing Alzheimer's disease. The investigators will conduct a randomized clinical trial with patients who have mild cognitive impairment (MCI). This is an early phase of memory loss that is worse than normal aging and may precede Alzheimer's disease. Patients will be randomized to either olfactory memory training or visual memory training for 3 months, with a final follow-up visit at 6 months. This study will attempt to determine if olfactory training is a useful for improving smell abilities, thinking abilities, and everyday functioning by examining change in these outcomes over time.

DETAILED DESCRIPTION:
There is an urgent and unmet need to develop interventions capable of improving cognition and everyday functioning in individuals at risk for cognitive decline. Olfactory training consists of systematic exposures to odors, with multiple reviews and meta-analyses concluding it has beneficial effects on cognition and olfaction. The application of olfactory training for preventing cognitive decline in MCI has received limited attention. The overarching goal of the research to be carried out in this application is to determine the feasibility and efficacy of Olfactory Memory Training (OMT) for patients with mild cognitive impairment (MCI). 30 patients with MCI will be recruited from the Memory Disorders Center at the New York State Psychiatric Institute and randomized to 3 months of OMT or active control training. OMT will involve an odor memory task, during which patients sample containers consisting of pairs of commercially available odors (flavored tea leaves). During each training session, non-descript containers are placed on a grid. On each trial, patients sample two containers, and attempt to find a match. The active control involves Visual Memory Training (VMT) with matching of abstract symbols rather than odors. Patients will complete 48 training sessions at home lasting approximately 10 minutes each. At baseline, 3 months, and 6 months follow-up, patients will complete a battery of cognitive, olfactory, and functional measures. In Aim 1, the investigators will compare change in cognitive (Preclinical Alzheimer Composite-5 [PACC5]) and olfactory functioning (Sniffin' Sticks Threshold, Discrimination, and Identification [TDI]) over 6 months in OMT versus VMT. In Aim 2, the investigators will compare change in everyday functioning (Alzheimer's Disease Cooperative Study-Activities of Daily Living scale - Prevention Instrument [ADCS-ADL-PI]) over 6 months in OMT versus VMT. If successful, this study has potential to develop a low-cost and scalable intervention. This study will inform the design of subsequent larger trials of OMT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-89 at the time of informed consent.
2. Montreal Cognitive Assessment score >=17.
3. Subjective cognitive complaints, i.e., memory or other cognitive complaints, e.g., naming/language.
4. Meets criteria for cognitive impairment (CI), including either early mild cognitive impairment (eMCI) or late mild cognitive impairment (lMCI), defined as memory function documented by scoring below the education adjusted cutoff on the Logical Memory II subscale (Story A, Delayed Paragraph Recall) from the Wechsler Memory Scale (WMS) - III (the maximum score is 25). The criteria for MCI (includes eMCI and lMCI) are as follows: eMCI is defined by a WMS-III Logical memory delayed recall score of 3-6 with 0-7 years of education, score of 5-9 with 8-15 years of education, and score of 9-11 with 16 or more years of education. lMCI is defined by a WMS-III Logical Memory delayed recall score ≤ 2 with 0-7 years of education, score ≤ 4 with 8-15 years of education, and score ≤ 8 with ≥ 16 years of education.
5. An informant (relative, friend, other caregiver) who contacts the participant at least weekly is required to provide information about the participant's functioning. If the informant drops out, an alternate informant can be designated by the participant.

Exclusion Criteria:

1. Diagnosis of dementia of any type.
2. Neurological disorders including Parkinson's disease, Huntington's disease, multiple sclerosis, stroke, epilepsy, traumatic brain injury (moderate to severe, with greater than 30 min loss of consciousness), and other neurologic disorders with focal signs (e.g., amyotrophic lateral sclerosis).
3. Current clinical diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, alcohol use disorder, or substance use disorder (Diagnostic and Statistical Manual of Mental Disorders (DSM)-5-Text Revision criteria).
4. Current unstable or untreated major depression, Geriatric Depression Scale (Short Form) score >= 6, or active suicidality based on a suicide scale (Columbia-Suicide Severity Rating Scale Screen version: positive answer to question 1 or 2 followed by item 6 positive answer leads to exclusion. Negative answer to questions 1 and 2: interview ends and the participant is not excluded for active suicidality).
5. Acute, severe unstable medical illness in the judgment of the clinician. For cancer, acutely ill participants (including those with metastases) are excluded, but history of successfully treated cancer does not result in exclusion.
6. Participation concurrently in another therapeutic clinical trial of a cognitive enhancing drug or device or procedure.
7. Current upper respiratory infection (participant rescheduled as soon as this improves), current smoker >1 pack daily (past smoking has been shown not to affect odor identification scores), self-reported congenital anosmia.
8. Severe vision, hearing, or tactile impairment that would prevent the participant from performing the cognitive tests accurately. This will be a clinical determination.
9. History of severe or recent asthma (defined as use of an inhaler for asthma, use of other asthma medication, or occurrence of an asthma attack within the last ten years), known special sensitivities to volatile chemicals, anyone who believes she is pregnant or is nursing a baby, and anyone who is on nasally administered medications other than people on nasal steroids to control rhinitis, allergic and otherwise.
10. Sino-nasal Outcome Test-22 nasal domain score >21, or individual score = 5, representing severe nasal symptoms that interfere with olfaction.
11. Allergies to any odors used in the olfactory testing or olfactory memory training.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Preclinical Alzheimer's Cognitive Composite 5 (PACC5) | Baseline, 3 Months, 6 Months
  The PACC5 provides a comprehensive assessment of Alzheimer's disease-relevant cognitive impairment and to serve as a tool with validated sensitivity to detect cognitive decline over time. It is comprised of five tests: Mini-Mental State Examination (total score range 0-30), Wechsler Memory Scale-Revised Logical Memory Delayed Recall (total score range 0-25), Digit-Symbol Coding Test (total score range 0-93), Free and Cued Selective Reminding Test Free + Total Recall (total score range 0-96), and Category Fluency Test (graded by number of correct words belonging in the categories of animals, fruits, and vegetables; not graded on a scale). The PACC5 is computed as an averaged z-score of all five tests.
Change in Sniffin' Sticks TDI (Threshold, Discrimination, and Identification composite) | Baseline, 3 Months, 6 Months
  The Sniffin' Sticks TDI test consists of a threshold test, a discrimination test, and an identification test. The results of the three subtests makes a total TDI score, where the minimum score is 1 and the maximum score is 48. A score >30 indicates normal olfactory function, a score between 15-30 indicates hyposmia and a score <15 indicates anosmia in the form of severely impaired or complete loss of olfaction.
Change in Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale (ADCS-ADL-PI) | Baseline, 3 Months, 6 Months
  The range of scores of the 15 items ADL question is 0-45 with higher scores indicating better daily functioning. This is the ADCS-ADL-PI outcome measure. In addition, there is a range of scores for the 5 items of physical function questions, which is 0-5 with higher scores indicating intact physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey N Motter, PhD, Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make de-identified data available to qualified users through a data repository (current plan is to use AD Knowledge Portal).
Supporting Information: SAP, ICF
Time Frame: The research community will have access to data starting 6 months after the publication of the results that address the Aims of the study.